CLINICAL TRIAL: NCT03061279
Title: Randomized Clinical Trial Evaluating Acutrak Headless Compression Screw Fixation of Medial Malleolus Fractures
Brief Title: Clinical Trial Evaluating Acutrak Headless Compression Screw Fixation of Medial Malleolus Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problem negotiating other sites
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Derek Amanatullah, Assistant Professor, Dept of Orthopedic Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37630
Record Dates: First submitted 2017-02-11; First posted 2017-02-23 (Actual); Results first posted 2020-03-02 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Medial Malleolus Fractures
Keywords: Medial Malleolus fractures; headless screws; headed screws
MeSH Terms: conditions — Ankle Fractures | interventions — Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fixation by Acutrak headless screw (Experimental)
  Interventions: Device: Fixation by Acutrak headless screw
- Fixation by headed screws, plates and or wire (Active Comparator): DePuy-Synthes Cannulated Cancellous Screws, DePuy-Synthes Cancellous Screws, DePuy-Synthes Cortical Screws, DePuy-Synthes 1/3 Tubular Plate, DePuy-Synthes LC-DCP Plate, DePuy-Synthes Pre-contoured Plate, and/or 18g Wire.
  Interventions: Device: Fixation by headed screws, plates, and or wires

INTERVENTIONS:
Device: Fixation by Acutrak headless screw — The fixation provided by the Acutrak headless compression screws provide sufficient fixation to achieve union and a favorable clinical outcome in both horizontal and vertical medial malleolus fractures when compared to bicortical and unicortical screw fixation, tension band wiring, and mini-fragment or buttress plating
  Other Names: Acutrak 2 Headless Compression Screw System
  Arms: Fixation by Acutrak headless screw
Device: Fixation by headed screws, plates, and or wires — DePuy-Synthes Cannulated Cancellous Screws, DePuy-Synthes Cancellous Screws, DePuy-Synthes Cortical Screws, DePuy-Synthes 1/3 Tubular Plate, DePuy-Synthes Locking contrast dynamic compression (LC-DCP) Plate, DePuy-Synthes Pre-contoured Plate, and/or 18g Wire are the alternative methods of treatment of medial malleolus fracture.
  Arms: Fixation by headed screws, plates and or wire

SUMMARY:
The purpose of this study is assess the safety and efficacy of Acutrak headless screws in comparison to other fixation methods (traditional headed screws, plates, and wires) used in the treatment of medial malleolus fracture of the ankle joint.

The investigators hope to learn the following objectives from this study

1. Prospectively establish equivalence with respect to fracture union rate after Acutrak headless compression screw fixation when compared to other fixation methods for medial malleolus fractures.
2. Prospectively establish equivalence with respect Patient Reported Outcome Measurement Information System (PROMIS) scores after Acutrak headless compression screw fixation when compared to other fixation methods for medial malleolus fractures.
3. Prospectively establish superiority with respect to hardware related pain after Acutrak headless compression screw fixation when compared to other fixation methods for medial malleolus fractures.
4. Prospectively establish superiority with respect to the hardware removal rate after Acutrak headless compression screw fixation when compared to other fixation methods for medial malleolus fractures.

Patients scheduled for open reduction and internal fixation for medial malleolus fracture by using Acutrak headless screw or any other method will be asked to enroll by the attending physician, and those patients will be asked to consent to the study. Patients will be randomized by sealed envelope to surgical fixation with traditional headed screws, plates, and wires or Acutrak headless compression screws. At the time of randomization, the fracture pattern and severity, past medical history and medications, and demographic data will be documented. After operative fixation, patients will receive routine fracture follow-up with a clinical evaluation for tenderness, radiographs to evaluate stability and union, and complete the PROMIS and Visual Analogue Pain Scale (VAS) scores to 2 weeks, 6 weeks, 3 months, 6 months, 1 year, and 2 years after surgical fixation

ELIGIBILITY:
Inclusion Criteria:

* Ankle fractures that undergo open reduction internal fixation of the medial malleolus

Exclusion Criteria:

* Tibial plafond (pilon) fractures
* Medial malleolar osteotomies to access the talus, perform an ankle fusion, or deal with a pathologic lesion, osteonecrosis, or infection due to their diversity in diagnosis, management, and weight bearing status
* Patients with prior surgical treatment of the ankle for fracture, deformity, infection, neoplasia, or other pathologic process on the ipsilateral extremity
* Patients that are non-weight bearing on one or both lower extremities prior to sustaining their ankle injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Amanatullah, MD, Study Director — Stanford University School of Medicine, CA; Micheal Weaver, MD, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School, Boston, MA; Domingo Hallare, MD, Principal Investigator — Kaiser Permanente Hospital, South Sacramento, CA
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Palo Alto, California
  - Kaiser Hospital, Sacramento, California
  - Brigham and Women's Hospital,, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rovinsky D, Haskell A, Liu Q, Paiement GD, Robinovitch S. Evaluation of a new method of small fragment fixation in a medial malleolus fracture model. J Orthop Trauma. 2000 Aug;14(6):420-5. doi: 10.1097/00005131-200008000-00007. PMID 11001416
- [Background] Toolan BC, Koval KJ, Kummer FJ, Sanders R, Zuckerman JD. Vertical shear fractures of the medial malleolus: a biomechanical study of five internal fixation techniques. Foot Ankle Int. 1994 Sep;15(9):483-9. doi: 10.1177/107110079401500905. PMID 7820240
- [Background] Amanatullah DF, McDonald E, Shellito A, Lafazan S, Cortes A, Curtiss S, Wolinsky PR. Effect of mini-fragment fixation on the stabilization of medial malleolus fractures. J Trauma Acute Care Surg. 2012 Apr;72(4):948-53. doi: 10.1097/TA.0b013e318249697d. PMID 22491610
- [Background] Amanatullah DF, Wolinsky PR. An alternative fixation technique for small medial malleolus fractures. Orthopedics. 2010 Dec;33(12):888. doi: 10.3928/01477447-20101021-17. No abstract available. PMID 21117562
- [Background] Dumigan RM, Bronson DG, Early JS. Analysis of fixation methods for vertical shear fractures of the medial malleolus. J Orthop Trauma. 2006 Nov-Dec;20(10):687-91. doi: 10.1097/01.bot.0000247075.17548.3a. PMID 17106379
- [Background] Amanatullah DF, Khan SN, Curtiss S, Wolinsky PR. Effect of divergent screw fixation in vertical medial malleolus fractures. J Trauma Acute Care Surg. 2012 Mar;72(3):751-4. doi: 10.1097/TA.0b013e31823b8b9f. PMID 22491565
- [Background] Brown OL, Dirschl DR, Obremskey WT. Incidence of hardware-related pain and its effect on functional outcomes after open reduction and internal fixation of ankle fractures. J Orthop Trauma. 2001 May;15(4):271-4. doi: 10.1097/00005131-200105000-00006. PMID 11371792
- [Background] Hung M, Baumhauer JF, Latt LD, Saltzman CL, SooHoo NF, Hunt KJ; National Orthopaedic Foot & Ankle Outcomes Research Network. Validation of PROMIS (R) Physical Function computerized adaptive tests for orthopaedic foot and ankle outcome research. Clin Orthop Relat Res. 2013 Nov;471(11):3466-74. doi: 10.1007/s11999-013-3097-1. PMID 23749433

RESULTS

PARTICIPANT FLOW:
Groups:
- Acutrak Fixation: Fixation by Acutrak headless screw: The fixation provided by the Acutrak headless compression screws provide sufficient fixation to achieve union and a favorable clinical outcome in both horizontal and vertical medial malleolus fractures when compared to bicortical and unicortical screw fixation, tension band wiring, and mini-fragment or buttress plating
- Standard of Care Fixation: Fixation by headed screws, plates, and or wires: DePuy-Synthes Cannulated Cancellous Screws, DePuy-Synthes Cancellous Screws, DePuy-Synthes Cortical Screws, DePuy-Synthes 1/3 Tubular Plate, DePuy-Synthes Locking contrast dynamic compression (LC-DCP) Plate, DePuy-Synthes Pre-contoured Plate, and/or 18g Wire are the alternative methods of treatment of medial malleolus fracture.
Period: Overall Study
Arm/Group | Acutrak Fixation | Standard of Care Fixation
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Acutrak fixation group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acutrak Fixation | Standard of Care Fixation | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Hardware Related Pain Localized to the Medial Malleolus at One Year After Sustaining an Ankle Fracture.
Description: Pain on a visual analogue scale (range: 0 to 1; 0 = no pain; 10 = worst pain imaginable).
Time Frame: Baseline, year 1
Population: No analysis was conducted due to small sample size and confidentiality concerns.
Arm/Group | Acutrak Fixation | Standard of Care Fixation
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Fracture Union Rate at One Year After Sustaining an Ankle Fracture.
Description: Fracture union rate assessed by radiographic imaging.
Time Frame: Month 3
Population: No analysis was conducted due to small sample size and confidentiality concerns.
Arm/Group | Acutrak Fixation | Standard of Care Fixation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Scores at Two Years After Sustaining an Ankle Fracture - Lower Extremity Function Scale (LEFS)
Description: The PROMIS LEFS scale consists of 20 questions, each on a 5-point Likert scale (0 = extreme difficulty, 4 = no difficulty). Questions are summed for a total score.
Time Frame: Baseline, year 2
Population: No analysis was conducted due to small sample size and confidentiality concerns.
Arm/Group | Acutrak Fixation | Standard of Care Fixation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Scores at Two Years After Sustaining an Ankle Fracture - Depression
Description: The PROMIS depression score is based on an adaptive test, and reported as a cumulative T-score with standard error.
Time Frame: Baseline, year 2
Population: No analysis was conducted due to small sample size and confidentiality concerns.
Arm/Group | Acutrak Fixation | Standard of Care Fixation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Scores at Two Years After Sustaining an Ankle Fracture - Pain Interference
Description: The PROMIS pain interference score is based on an adaptive test, and reported as a cumulative T-score with standard error.
Time Frame: Baseline, year 2
Population: No analysis was conducted due to small sample size and confidentiality concerns.
Arm/Group | Acutrak Fixation | Standard of Care Fixation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Scores at Two Years After Sustaining an Ankle Fracture - Physical Function
Description: The PROMIS physical function score is based on an adaptive test, and reported as a cumulative T-score with standard error.
Time Frame: Baseline, year 2
Population: No analysis was conducted due to small sample size and confidentiality concerns.
Arm/Group | Acutrak Fixation | Standard of Care Fixation
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Amount Pain Medication Required During Recovery Period
Description: Pain medication measured in morphine equivalents.
Time Frame: Up to 2 years
Population: No analysis was conducted due to small sample size and confidentiality concerns.
Arm/Group | Acutrak Fixation | Standard of Care Fixation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Plan was to follow adverse events for up to 2 years.
Description: No participants were enrolled in the Acutrak Fixation group.
Arm/Group | Acutrak Fixation | Standard of Care Fixation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT03061279/Prot_SAP_000.pdf